CLINICAL TRIAL: NCT06388980
Title: Knowledge and Needs of Nursing Professionals in Relation to the Treatment of People With Complex Wounds at Parc Taulí University Hospital
Brief Title: Knowledge and Needs of Nursing in Relation to the Treatment Complex Wounds
Status: Active, not recruiting | Type: Observational
Sponsor: Corporacion Parc Tauli (Other)
Responsible Party: Principal Investigator, Francisco Zamora Carmona, Advanced Practice Wound Nurse, Corporacion Parc Tauli
Other Study IDs: UFCIN1_2022
Record Dates: First submitted 2024-04-18; First posted 2024-04-29 (Actual); Last update posted 2025-02-20 (Actual); Status verified 2025-02

CONDITIONS: Nurse's Role; Knowledge, Attitudes, Practice; Wound
Keywords: nurses; complex wounds; knowledge
MeSH Terms: conditions — Behavior; Wounds and Injuries

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Prospective
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

INTERVENTIONS:
Other: Validated questionnaires and ad hoc questions — validated questionnaires and open questions online through the institution's intranet anonymous
  Other Names: validated questionnaires and open questions

SUMMARY:
Study with cross-sectional and descriptive mixed methodology. With questionnaires with likert-type questions (0-10) being the 10 with the highest score, and open questions in relation to knowledge in wound care; include all Corporaciló Sanitària Parc Taulí (CCSPT) nurses who voluntarily want to participate in a pseudo-anonymized surv

DETAILED DESCRIPTION:
INTRODUCTION A complex wound is a skin injury with little or no tendency to heal as long as the cause that produces it is present. Complex wounds that are difficult to heal or develop torpid or refractory to the usual treatments, do not evolve adequately in the expected time (> 6 weeks).

The clinical practice we find is completely heterogeneous among professionals who care for people with injuries.

OBJECTS Describe the knowledge and training needs perceived by nurses in the approach to people with complex wounds of the CCSPT.

To explore the difficulties and facilitating elements that professionals perceive when dealing with people with complex wounds, from the reference area of the Parc Taulí University Hospital, over a period of 12 months.

Explain tools with scientific evidence for correct continuity of care.

METHODOLOGY:

Study with cross-sectional and descriptive mixed methodology. With questionnaires with likert-type questions and open questions in relation to knowledge in wound care; include all CCSPT nurses who voluntarily want to participate in a pseudo-anonymized survey.

EXPECTED RESULTS:

Current situation of the knowledge, needs, limiting and facilitating elements that nursing professionals have to address people with injuries.

ELIGIBILITY:
Inclusion Criteria:

* Nurses who take care of people with both adult and pediatric injuries.
* Nurses who give their informed consent to participate in the study voluntarily.

Exclusion Criteria:

* Nurses who do not want to participate in the study voluntarily.
* Nurses who do not have healthcare activities (due to workplace, due to long-term illness, absence from work)

Sex: All
Age Groups: Child, Adult, Older Adult
Study Population: Acute and social healthcare hospital nurses
Sampling Method: Non-Probability Sample
Enrollment: 200 (Estimated)
Dates: Start 2023-05-01 (Actual); Primary Completion 2023-06-01 (Actual); Study Completion 2028-06-01 (Estimated)

PRIMARY OUTCOMES:
"What not to do in chronic wounds?" | 1 month
  made up of socio-demographic variables of the participants: gender, age, level of education, years working as a nurse, training on wounds. And 37 items with three answer options "true", "fake" in relation to the 37 recommendations of the document "What not to do in chronic wounds?", the more correct, the more knowledge about wounds.
ReAc-PUKT (Renobato-Acosta Pressure Ulcer Knowledge Test) | 1 month
  To determine knowledge of nurses about the prevention and treatment of pressure injuries (LPP). The instrument is made up of two sections: The first collects general data on professionals and academic-work information, including socio-demographic data (age, gender), service to which they belong, work shift, years of experience, academic training and training in LPP. The second measures the level of scientific knowledge about pressure injuries) generalities, prevention and treatment, the more correct, the more knowledge about LPP. The higher the value, the better the knowledge about LPP.

SECONDARY OUTCOMES:
Ad hoc open questions | 1 month
  Researchers want to know the training needs perceived by nursing staff and the limiting and facilitating elements they experience in dealing with people with complex injuries.
  The qualitative methodology of descriptive phenomenological approach, through 10 open questions that will give us relevant information for the study:
  * Learn about their experiences in care.
  * Learn about their experiences with people with injuries.
  * Explore the difficulties and facilitating elements when making referrals and interconsultations with specialists.
  * Explain the tools we have with scientific evidence for correct continuity of care
  * Know the facilitating elements in the continuity of care.

CONTACTS AND LOCATIONS:
Overall Officials: Francisco Zamora Carmona, Principal Investigator — Grupo emergente enfermeria I3PT
Locations (1):
- Corporació Sanitària Parc Taulí, Sabadell, Barcelona, Spain

IPD SHARING:
Plan to Share IPD: No